CLINICAL TRIAL: NCT05558098
Title: Dapagliflozin in Patients With Critical Illness: A Randomized Controlled Trial
Brief Title: Dapagliflozin in Patients With Critical Illness
Acronym: DEFENDER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEFENDER
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Critical Illness; Sepsis
Keywords: dapagliflozin; critical illness
MeSH Terms: conditions — Critical Illness; Sepsis | interventions — dapagliflozin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Current standard of care for critically ill patients.
  Interventions: Other: Standard of Care
- Standard of care plus dapagliflozin (Active Comparator): Current standard of care for critically ill patients plus open-label dapagliflozin 10 mg per day for 14 days or until ICU discharge
  Interventions: Drug: Dapagliflozin 10mg Tab

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin 10 mg once per day for 14 days or until intensive care unit discharge or death
  Other Names: Farxiga
  Arms: Standard of care plus dapagliflozin
Other: Standard of Care — Current standard of care for management of critically ill patients
  Arms: Standard of Care

SUMMARY:
To assess the effects of dapagliflozin on a composite hierarchical endpoint in critically ill patients.

DETAILED DESCRIPTION:
Critically ill patients in the intensive care unit (ICU) experience a high mortality rate. Recent data indicates that the mortality rate for unplanned ICU admissions exceeds 30%, highlighting the urgent need for therapies that can reduce mortality in these critical patients.

DEFENDER is an investigator-initiated, multi-center, randomized, open-label clinical trial, conducted in Brazilian ICUs.

The study population will consist of participants who have been admitted to an ICU with an expected length of stay of more than 48 hours with evidence of at least an acute organ dysfunction, such as hypotension, signs of acute kidney injury, and/or the need for new use of high-flow nasal catheter, noninvasive or invasive ventilation. Eligible patients will be enrolled within 24 hours after the onset of organ dysfunction.

Participants will be randomly assigned in a 1:1 ratio to receive either dapagliflozin 10mg (for 14 days or until ICU discharge, whichever occurs sooner) in addition to standard of care, or standard care alone.

The primary outcome of the study is a hierarchical composite endpoint, including: i) hospital mortality, ii) initiation of kidney-replacement therapy, and iii) ICU length of stay. These outcomes will be assessed up to 28 days after randomization, with censoring at the time of hospital discharge.

To ensure participant safety, an independent Data and Safety Monitoring Board will periodically review the data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to an intensive care unit with expected duration of admission of at least 48 hours in the opinion of the attending physician AND
2. Patients with at least one new organ dysfunction:

   1. Hypotension (mean arteria pressure below 65 mmHg or systolic blood pressure below 90 mmHg or use of vasopressors - norepinephrine, epinephrine, adrenaline, or vasopressin at any dose);
   2. Signs of acute kidney injury (increase in serum creatinine above 0.3 mg/dL over previous measurement or decrease in urinary output - below 0.5 mL/kg/h - in the past six hours;
   3. Need for new use of high-flow nasal catheter or noninvasive ventilation or invasive ventilation.

Exclusion Criteria:

1. Pregnancy or age below 18 years;
2. Patient or legal representative refusal;
3. Patients with chronic kidney disease on dialysis;
4. Planned intensive care unit admission after elective surgery;
5. Known allergy to dapagliflozin;
6. Previous use of dapagliflozin or other sodium-glucose transport protein 2 inhibitor;
7. Patients that cannot receive medications through oral or enteral route;
8. Patients with inclusion criteria number 2 for more than 24 hours.
9. Patients with type 1 diabetes or previous ketoacidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Win Ratio | 28 days
  Hierarchical endpoint of hospital mortality, use of kidney replacement therapy and intensive care unit length-of-stay

SECONDARY OUTCOMES:
Hospital Mortality | 28 days
  Death within index hospitalization
Use of kidney replacement therapy | 28 days
  Use of kidney replacement therapy during hospital stay
Intensive Care Unit Free Days | 28 days
  Number of days patient was alive and not in the intensive care unit within index hospitalization
Hospital Free Days | 28 days
  Number of days patient was alive and not in the hospital
Vasopressor Free Days | 28 days
  Number of days patient was alive and not using vasopressors at any dose within index hospitalization
Mechanical Ventilation Free Days | 28 days
  Number of days patient was alive and not using mechanical ventilation within index hospitalization
Kidney Replacement Therapy Free Days | 28 days
  Number of days patient was alive and not using kidney replacement therapy within index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Otavio Berwanger, PhD, Study Chair — Academic Research Organization
Locations (23):
- Brazil (23):
  - Hospital de Emergência Dr. Daniel Houly, Arapiraca, Alagoas
  - Hospital e Maternidade São José, Colatina, Espírito Santo
  - Instituto de Ensino e Pesquisa do Hospital da Bahia, Salvador, Estado de Bahia
  - Hospital Brasilia, Brasília, Federal District
  - Hospital Municipal de Aparecida de Goiânia, Aparecida de Goiânia, Goiás
  - Hospital Santa Lucia, Poços de Caldas, Minas Gerais
  - Hospital das Nações, Curitiba, Paraná
  - Hospital Ecoville - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital Nossa Senhora da Oliveira, Vacaria, Rio Grande do Sul
  - Hospital Baia Sul, Florianópolis, Santa Catarina
  - Centro de Pesquisa Clínica do Coração, Aracaju, Sergipe
  - Hospital de Amor de Barretos, Barretos, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Nove de Julho, São Paulo, São Paulo
  - Santa Casa de Barretos, Barretos
  - Santa Casa de Curitiba, Curitiba
  - Hospital de Amor de Jales, Jales
  - Unimed Joinville, Joinville
  - Hospital São Lucas de Copacabana, Rio de Janeiro
  - Hospital Municipal Vila Santa Catarina, São Paulo
  - Hospital M´Boi Mirim, São Paulo
  - Hospital Santa Paula, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonable request after approval of the steering committee

REFERENCES:
- [Derived] Tavares CAM, Azevedo LCP, Guimaraes PO, Rea-Neto A, David-Joao PG, Campos NS, Amendola CP, Kozesinski-Nakatani AC, Filiponi TC, Almeida GMB, Bergo RR, Lobo SM, Tognon AP, Tavares MS, Silveira FS, Dracoulakis MDA, Biondi RS, Monfardini F, Nieri J, Madrini V Jr, Serpa-Neto A, Bacal F, Lemos PA, Berwanger O, Ezekowitz JA, Zampieri FG; DEFENDER Investigators. Dapagliflozin in Acute Cardiovascular Conditions: Insights From the DEFENDER Trial. JACC Adv. 2025 Dec 19;5(1):102459. doi: 10.1016/j.jacadv.2025.102459. Online ahead of print. PMID 41421016
- [Derived] Tavares CAM, Azevedo LCP, Rea-Neto A, Campos NS, Amendola CP, Kozesinski-Nakatani AC, David-Joao PG, Lobo SM, Filiponi TC, Almeida GMB, Bergo RR, Guimaraes-Junior MRR, Figueiredo RC, Castro JR, Schuler CJ, Westphal GA, Carioca ACR, Monfradini F, Nieri J, Neves FMO, Paulo JA, Albuquerque CSN, Silva MCR, Kosiborod MN, Pereira AJ, Damiani LP, Correa TD, Serpa-Neto A, Berwanger O, Zampieri FG; DEFENDER Investigators. Dapagliflozin for Critically Ill Patients With Acute Organ Dysfunction: The DEFENDER Randomized Clinical Trial. JAMA. 2024 Aug 6;332(5):401-411. doi: 10.1001/jama.2024.10510. PMID 38873723
- [Derived] Tavares CAM, Azevedo LCP, Rea-Neto A, Campos NS, Amendola CP, Bergo RR, Kozesinski-Nakatani AC, David-Joao PG, Westphal GA, Guimaraes Junior MRR, Lobo SMA, Tavares MS, Dracoulakis MDA, Souza GM, Almeida GMB, Gebara OCE, Tomba PO, Albuquerque CSN, Silva MCR, Pereira AJ, Damiani LP, Correa TD, Serpa-Neto A, Berwanger O, Zampieri FG. Dapagliflozin in patients with critical illness: rationale and design of the DEFENDER study. Crit Care Sci. 2023 Dec 22;35(3):256-265. doi: 10.5935/2965-2774.20230129-en. eCollection 2023. PMID 38133155